CLINICAL TRIAL: NCT01192477
Title: Ozone Cardiovascular Effects in Genetically Susceptible People
Acronym: OZCARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH); Conservation of Clean Air and Water in Europe (CONCAWE) (Unknown); Exxon Mobil (Industry)
Responsible Party: Principal Investigator, Mark Frampton, Professor, University of Rochester
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 017428; R01ES017428-01A1 (NIH)
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
Keywords: Air pollution; Ozone; Health effects of ozone exposure
MeSH Terms: interventions — Ozone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ozone 0.1 ppm (Experimental)
  Interventions: Other: Ozone
- Ozone 0.2 ppm (Experimental)
  Interventions: Other: Ozone
- Filtered air (Sham Comparator)
  Interventions: Other: Ozone

INTERVENTIONS:
Other: Ozone — All subjects will have a 3-hour exposure to clean air, a 3-hour exposure to clean air with lower ozone (0.1 ppm), and a 3-hour exposure to clean air with higher ozone (0.2 ppm). Exposures will take place at least 3 weeks apart. Order of exposure will be randomized for each subject.
  Other Names: Ozone exposure; Ozone air pollution

SUMMARY:
Increases in air pollution are associated with increases in deaths from cardiovascular disease, but the investigators know little about how ozone air pollution affects the cardiovascular system. The investigators proposed study will determine the effects of ozone on blood vessel and heart function that could worsen illness in people with underlying heart disease. This will be accomplished by studying healthy volunteers who inhale ozone in a controlled clinical study, and also by studying their exposure to ozone and other pollutants during their normal daily activities. The investigators will study volunteers who may be at increased risk for the effects of ozone because of genetic susceptibility. Understanding the effects of ozone on the heart and circulation can help establish appropriate air pollution standards, and provide strategies to protect the most susceptible people.

ELIGIBILITY:
Inclusion Criteria:

* Healthy,
* Never-smokers with normal spirometry based on the standards published by Morris and co-workers (Morris et al. 1971), and
* A normal electrocardiogram. -

Exclusion Criteria:

* Any history of habitual smoking.
* Marijuana smoking within the past 5 years.
* Pregnancy.
* Any history of significant organ impairment, chronic respiratory disease, ischemic heart disease, active psychiatric disorder or current drug or alcohol abuse.
* Occupation involving regular, heavy dust or particle exposure, such as welding, mining, foundry work.
* FEV1 < 75% of predicted at baseline screening.
* Subjects with atopy or allergic rhinitis will not be excluded as long as they do not require regular treatment with antihistamines or systemic steroids.
* Subjects on certain prescription medications such as prednisone or statins will be excluded. Use of other medications will be considered on an individual basis. Subjects will not be asked to discontinue prescription medications for the purposes of this study.
* Hypertension (blood pressure higher than 140/90 mmHg or on antihypertensive medication).
* Subject lives outside the Rochester metropolitan area.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Nitric oxide bioavailability | Before and 3 hours after ozone exposure
  We hypothesize that systemic vascular effects of exposure to ozone will be reflected in reductions in arterial blood nitrite or its A/V gradient. This will require simultaneous collection of venous and arterial blood.

SECONDARY OUTCOMES:
Evidence of endothelial injury | Before and 3 hours after ozone exposure
  We hypothesize that systemic vascular effects of exposure to ozone will alter markers of vascular function and inflammation. Flow cytometry will be used to detect activated platelets and pro-coagulant circulating microparticles.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Frampton, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States